CLINICAL TRIAL: NCT02883673
Title: Prospective, Single Arm Pivotal Clinical Trial Designed to Assess the Safety and Effectiveness of the Jada System in Treating Primary Postpartum Hemorrhage
Brief Title: Safety and Effectiveness of the Jada System in Treating Primary Postpartum Hemorrhage
Acronym: PEARLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alydia Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-01 v2.6; PPH-02 (Other: Alydia Health)
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Results first posted 2022-04-12 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Postpartum Hemorrhage
Keywords: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Intervention (Experimental): Jada System for Postpartum Hemorrhage will be administered to subjects who are diagnosed with postpartum hemorrhage.
  Interventions: Device: Jada System

INTERVENTIONS:
Device: Jada System — It is a teardrop-shaped, soft silicone ring that is placed into the uterus, where gentle suction is applied to cause the uterus to contract and shrink in size, compressing the blood vessels so the bleeding stops.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Jada System in the control and reduction of primary postpartum hemorrhage.

DETAILED DESCRIPTION:
This IDE study is designed to evaluate the effectiveness and safety of the Jada System to treat primary PPH. The study is literature controlled.

ELIGIBILITY:
Inclusion Criteria:

1. Adult Female, 18 years of age or older at time of consent.
2. Able to understand and provide informed consent to participate in the study.
3. Diagnosis of PPH with suspected atony within 24 hours after vaginal or c-section delivery.
4. EBL, to be determined when investigator is ready to have Jada peel pack opened: a) vaginal delivery: 500 - 1500 ml EBL or b) c-section delivery: 1000 - 1500 ml EBL.
5. Failed first-line intervention of uterotonics and uterine massage/bimanual compression to stop bleeding. Note: Uterotonic administration may continue concomitant with and post Jada use.

Exclusion Criteria:

1. EBL > 1500 ml, to be determined when investigator is ready to have the Jada peel pack opened.
2. Delivery at a gestational age < 34 weeks.
3. For C-sections: Cervix < 3 cm dilated before Jada use.
4. PPH that the investigator determines to require more aggressive treatment, including any of the following: a) hysterectomy, b) b-lynch suture, c) uterine artery embolization or ligation, d) hypogastric ligation.
5. Known uterine anomaly.
6. Ongoing intrauterine pregnancy.
7. Placenta abnormality including any of the following: a) known placenta accreta, b) retained placenta with known risk factors for placenta accreta (e.g. history of prior uterine surgery, including prior c-section and placenta previa), c) retained placenta without easy manual removal.
8. Known uterine rupture.
9. Unresolved uterine inversion.
10. Subject has undergone intrauterine balloon therapy or uterine packing for tamponade treatment of this PPH prior to use of the Jada.
11. Current cervical cancer.
12. Current purulent infection of the vagina, cervix, uterus.
13. Diagnosis of coagulopathy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2017-09-17 (Actual); Primary Completion 2020-01-26 (Actual); Study Completion 2020-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary D'Alton, MD, Principal Investigator — Columbia University
Locations (15):
- United States (15):
  - University of Alabama Birmingham, Birmingham, Alabama
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - New York Presbyterian Queens, Flushing, New York
  - Nyph/Cumc, New York, New York
  - MetroHealth Case Western, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - UPMC - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - UT Health Science Center, McGovern School of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carroli G, Cuesta C, Abalos E, Gulmezoglu AM. Epidemiology of postpartum haemorrhage: a systematic review. Best Pract Res Clin Obstet Gynaecol. 2008 Dec;22(6):999-1012. doi: 10.1016/j.bpobgyn.2008.08.004. Epub 2008 Sep 25. PMID 18819848
- [Background] Khan KS, Wojdyla D, Say L, Gulmezoglu AM, Van Look PF. WHO analysis of causes of maternal death: a systematic review. Lancet. 2006 Apr 1;367(9516):1066-1074. doi: 10.1016/S0140-6736(06)68397-9. PMID 16581405
- [Background] McLintock C, James AH. Obstetric hemorrhage. J Thromb Haemost. 2011 Aug;9(8):1441-51. doi: 10.1111/j.1538-7836.2011.04398.x. PMID 21668737
- [Background] American College of Obstetricians and Gynecologists. ACOG Practice Bulletin: Clinical Management Guidelines for Obstetrician-Gynecologists Number 76, October 2006: postpartum hemorrhage. Obstet Gynecol. 2006 Oct;108(4):1039-47. doi: 10.1097/00006250-200610000-00046. PMID 17012482
- [Background] Schorn MN. Measurement of blood loss: review of the literature. J Midwifery Womens Health. 2010 Jan-Feb;55(1):20-7. doi: 10.1016/j.jmwh.2009.02.014. PMID 20129226
- [Background] Sapadin AN, Lebwohl MG, Teich SA, Phelps RG, DiCostanzo D, Cohen SR. Periumbilical pseudoxanthoma elasticum associated with chronic renal failure and angioid streaks--apparent regression with hemodialysis. J Am Acad Dermatol. 1998 Aug;39(2 Pt 2):338-44. doi: 10.1016/s0190-9622(98)70385-8. PMID 9703148
- [Background] Al-Zirqi I, Vangen S, Forsen L, Stray-Pedersen B. Prevalence and risk factors of severe obstetric haemorrhage. BJOG. 2008 Sep;115(10):1265-72. doi: 10.1111/j.1471-0528.2008.01859.x. PMID 18715412
- [Derived] Goffman D, Rood KM, Bianco A, Biggio JR, Dietz P, Drake K, Heilman E, Hopkins M, De Four Jones M, Katz T, Martin C, Prasad M, Smid MC, Wine KD, Ryan R, Yong C, Carney PI, Simhan HN. Real-World Utilization of an Intrauterine, Vacuum-Induced, Hemorrhage-Control Device. Obstet Gynecol. 2023 Nov 1;142(5):1006-1016. doi: 10.1097/AOG.0000000000005366. Epub 2023 Sep 13. PMID 37713322
- [Derived] D'Alton ME, Rood KM, Smid MC, Simhan HN, Skupski DW, Subramaniam A, Gibson KS, Rosen T, Clark SM, Dudley D, Iqbal SN, Paglia MJ, Duzyj CM, Chien EK, Gibbins KJ, Wine KD, Bentum NAA, Kominiarek MA, Tuuli MG, Goffman D. Intrauterine Vacuum-Induced Hemorrhage-Control Device for Rapid Treatment of Postpartum Hemorrhage. Obstet Gynecol. 2020 Nov;136(5):882-891. doi: 10.1097/AOG.0000000000004138. PMID 32909970

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 107
Completed | 107
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Jada Arm: Treatment Arm
Arm/Group | Jada Arm
Number analyzed (Participants) | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (5.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 88
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 61
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 107

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Rate of Participants With Cessation of Uterine Hemorrhaging
Description: Control of postpartum hemorrhage, defined as the avoidance of non-surgical, second-line or surgical intervention to control uterine hemorrhage after the use of the Jada System per the Instructions for Use
Time Frame: 24 hrs
Population: Group of participants for whom Jada was activated
Measure: Count of Participants; unit: Participants
Groups:
- ITT Population: Group where Jada treatment was applied
Arm/Group | ITT Population
Number analyzed (Participants) | 106
Participants | 100

2. Primary Outcome: Safety: Incidence (i.e., Rate or Number of Participants), Severity and Seriousness of Device-related Adverse Events Experienced by Participants
Description: Incidence (i.e., rate or number of participants), severity and seriousness of device-related Adverse Events experienced by participants will be documented during the course of the study.
Time Frame: 6 weeks
Population: Participants in whom Jada was activated
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 106
Participants | 8

ADVERSE EVENTS:
Time Frame: Adverse events were collected from patient admission through 6-week follow-up visit post discharge (follow-up visit window was 42 days +/- 14 days).
Description: Safety/Intent to Treat (ITT) Cohort: All subjects in whom treatment was attempted with Jada (i.e., device inserted, and vacuum turned on) were included in the Safety/ITT Cohort.
  One subject was excluded from the Safety/ITT analysis population as the Jada System was unable to be inserted and therefore vacuum treatment was not turned on/connected, leaving 106 subjects for the Safety/ITT Cohort. Notably there were no adverse events reported for this one excluded subject.
Arm/Group | ITT Population
All-Cause Mortality (participants affected / at risk) | 0/106
Serious Adverse Events (participants affected / at risk) | 18/106
Other Adverse Events (participants affected / at risk) | 45/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITT Population (N=106)
Endometritis (Infections and infestations) | 3 (3) — Endometritis
Anemia (Blood and lymphatic system disorders) | 3 (3) — Anemia
Anemia leading to hysterectomy (Blood and lymphatic system disorders) | 1 (1) — Anemia leading to hysterectomy
Anemia and tachycardia and hypotension (Blood and lymphatic system disorders) | 1 (1) — Anemia and tachycardia and hypotension
Continued bleeding due to undiscovered retained placenta (Blood and lymphatic system disorders) | 1 (1) — Continued bleeding due to undiscovered retained placenta
Hypotension with complaint of dyspnea and nausea (Cardiac disorders) | 1 (1) — Hypotension with complaint of dyspnea and nausea
Pregnancy related hypertension (Cardiac disorders) | 1 (1) — Pregnancy related hypertension
C-section incision repair bleed (Surgical and medical procedures) | 1 (1) — C-section incision repair bleed
Constipation and hemorrhoid (Gastrointestinal disorders) | 1 (1) — Constipation and hemorrhoid
Laceration of cervix during difficult amniotomy (Skin and subcutaneous tissue disorders) | 1 (1) — Laceration of cervix during difficult amniotomy
Acute tubular necrosis (Renal and urinary disorders) | 3 (3) — Acute tubular necrosis
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pulmonary edema
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Shortness of breath
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ITT Population (N=106)
Anemia (Blood and lymphatic system disorders) | 15 (15) — Anemia
Anemia with tachycardia (Blood and lymphatic system disorders) | 1 (1) — Anemia with tachycardia
Lower uterine segment clot requiring removal (Blood and lymphatic system disorders) | 1 (1) — Lower uterine segment clot requiring removal
Passed clots at 4 weeks postpartum with pain (Blood and lymphatic system disorders) | 1 (1) — Passed clots at 4 weeks postpartum with pain
Pretibial edema (Blood and lymphatic system disorders) | 1 (1) — Pretibial edema
Chest pain, SOB, diplopia, nausea without lab evidence of MI resolved without sequalae (Cardiac disorders) | 1 (1) — Chest pain, SOB, diplopia, nausea without lab evidence of MI resolved without sequalae
Pregnancy related hypertension (Cardiac disorders) | 2 (2) — Pregnancy related hypertension
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) — Cellulitis
Cellulitis with yeast (Skin and subcutaneous tissue disorders) | 1 (1) — Cellulitis with yeast
labial cyst (Skin and subcutaneous tissue disorders) | 2 (2) — labial cyst
Leg rash associated with medication for hypertension (Skin and subcutaneous tissue disorders) | 1 (1) — Leg rash associated with medication for hypertension
Constipation (Gastrointestinal disorders) | 2 (2) — Constipation
Dyspepsia (Gastrointestinal disorders) | 1 (1) — Dyspepsia
Hemorrhoid (Gastrointestinal disorders) | 1 (1) — Hemorrhoid
Presumed endometritis (Infections and infestations) | 1 (1) — Presumed endometritis
Presumed endometritis with pre-existing chorioamnionitis (Infections and infestations) | 1 (1) — Presumed endometritis with pre-existing chorioamnionitis
upper respiratory tract influenza (Infections and infestations) | 1 (1) — upper respiratory tract influenza
Presumed endometritis with leukocytosis (Infections and infestations) | 1 (1) — Presumed endometritis with leukocytosis
bacterial vaginosis (Infections and infestations) | 1 (1) — bacterial vaginosis
Chlamydia (Infections and infestations) | 1 (1) — Chlamydia
Endometritis (Infections and infestations) | 1 (1) — Endometritis
Mastitis (Infections and infestations) | 1 (1) — Mastitis
Uncomplicated urinary tract infection (Infections and infestations) | 2 (2) — Uncomplicated urinary tract infection
Vaginal yeast (Infections and infestations) | 1 (1) — Vaginal yeast
Migraine headache (Nervous system disorders) | 1 (1) — Migraine headache
Spinal headache (Nervous system disorders) | 1 (1) — Spinal headache
Vaginal pain and light bleeding from pre-existing laceration (Skin and subcutaneous tissue disorders) | 1 (1) — Vaginal pain and light bleeding from pre-existing laceration
Breast rash (Skin and subcutaneous tissue disorders) | 1 (1) — Breast rash
Breast pain possibly blocked duct (Reproductive system and breast disorders) | 1 (1) — Breast pain possibly blocked duct
Dysuria (Renal and urinary disorders) | 1 (1) — Dysuria
Headache (Nervous system disorders) | 1 (1) — Headache
Pelvic and perineal pain (Reproductive system and breast disorders) | 1 (1) — Pelvic and perineal pain
Anxiety (Psychiatric disorders) | 2 (2) — Anxiety
Depression (Psychiatric disorders) | 2 (2) — Depression
Depression, anxiety, PTSD (Psychiatric disorders) | 1 (1) — Depression, anxiety, PTSD
acute tubular necrosis (Renal and urinary disorders) | 1 (1) — acute tubular necrosis
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Hypoxia
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pulmonary edema
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Shortness of breath
Disruption of laceration repair (Skin and subcutaneous tissue disorders) | 1 (1) — Disruption of laceration repair

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT02883673/Prot_SAP_000.pdf